CLINICAL TRIAL: NCT05499611
Title: Contribution of Optical Genome Mapping to the Prognostic Classification of Acute Myeloblastic Leukemia Evaluation of the Clinical Utility of DNA Optical Mapping in the Management of Acute Myeloblastic Leukemia (COALA)
Brief Title: Impact of Optical Genome Mapping in Acute Myeloblastic Leukemia
Acronym: COALA
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/28
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloblastic Leukemia
Keywords: Optical Genome Mapping (OGM); Acute Myeloblastic Leukemia (AML); Complex Karyotype; Prognosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study using a new technology will be performed: the Optical Genome Mapping (OGM) on acute myelogenous leukemia (AML) samples stored at the CRB-Cancer of the Bordeaux University Hospital and annotated in the DATAML clinical database. The main objective is to estimate the proportion of AML patients for whom OGM detects at least one additional abnormality compared to conventional techniques. This study will constitute an important step in the validation of COA as a reference technique for cytogenetic analysis in AML, replacing the classical techniques, and could also constitute a first argument for redesigning the prognostic classification of AML.

DETAILED DESCRIPTION:
In AML prognostic classifications, such as the ELN 2017 classification, which are used to guide treatment choices in the majority of protocols, rely heavily on genetic abnormalities. The Optical Genome Mapping (OGM) is a new technology that combines in one and the same technique the results of karyotype, FISH and SNP-Array, the latter being very little used in current practice in AML. OGM with greater sensitivity and a better resolution than the usual techniques should therefore allow us to identify more abnormalities than conventional cytogenetics; we would then like to determine whether these additional abnormalities have a prognostic impact, i.e., whether they lead to reclassification of patients initially classified as "favorable" or "intermediate" into the "unfavorable" prognostic category, with therapeutic consequences.

A retrospective study using the OGM is will be performed on samples stored at the CRB-Cancer of the Bordeaux University Hospital and annotated in the DATAML clinical database. In an original way, the focus will be on AML patients in whom 1 to 3 chromosomal abnormalities (non-recurrent WHO, not related to an unfavourable prognosis) have already been demonstrated by classical techniques, making the hypothesis that it is in this population that we would more easily have patients who could fall into the definition of the complex karyotype and thus into the unfavourable risk category.

OGM should therefore reveal a greater number of abnormalities which would allow a better definition of karyotypes with abnormalities, the number of complex and/or monosomal karyotypes and a better stratification of the prognosis of these patients with AML. This is an applied translational research study based on innovative technology that will define the place of OGM over current techniques used in the initial management of AML patients, and it may well become the new standard for cytogenetic analysis of AML in the coming years.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years and ≤ 65 years of age who have been treated with intensive chemotherapy
* Diagnosis of AML (with a minimum follow-up of 24 months)
* Presence of samples included in CRB-K in the AML collection
* Cytogenetic data available: karyotype with 1-3 abnormalities present in one or more clones, excluding recurrent WHO abnormalities (t(8;21), inv(16) or t(16;16), t(9;11), t(v;11)(v;q23. 3), t(6;9), inv(3) or t(3;3) and t(9;22)) or assigned by itself to an unfavorable prognosis: -5 or del(5q); -7; -17/abn(17p).
* Molecular data available for the following genes: ASXL1, CEBPA, FLT3-ITD, NPM1, RUNX1 and TP53 (the list of genes of interest may be adapted according to the upcoming ELN 2022 classification)

Exclusion Criteria:

* Samples not included in the CRB-K (lack of consent, insufficient material...)
* Karyotype with one of the following abnormalities: (t(8;21), inv(16) or t(16;16), t(9;11), t(v;11)(v;q23.3), t(6;9), inv(3) or t(3;3), and t(9;22)) or associated with an unfavorable prognosis on its own: -5 or del(5q); -7; -17/abn(17p)
* Karyotype without clonal abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of AML (with a minimum follow-up of 24 months)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with more abnormalities detected by OGM than by conventional cytogenetics | At baseline

SECONDARY OUTCOMES:
Average number of additional abnormalities detected by OGM compared to conventional techniques | At baseline
Proportion of patients reclassified as complex and/or monosomal karyotype according to current ELN definitions | At baseline
Proportion of patients for whom a change in therapeutic management could have been proposed | From baseline to Month 36
Comparison of overall survival and event-free survival curves of patients reclassified to the unfavorable group to those of the intermediate and unfavorable groups in a historical cohort | From baseline to Month 36
Interobserver reproducibility for interpretation of OGM results (Fleiss Kappa coefficient) | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, service Hématologie Biologique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No